CLINICAL TRIAL: NCT03144986
Title: A Pilot Study to Determine the Safety and Efficacy of H-Coil Deep Transmagnetic Stimulation in Treatment Resistant Anorexia Nervosa
Brief Title: Insula-coil Deep TMS for Treatment Resistant Anorexia Nervosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Brainsway (Industry)
Responsible Party: Principal Investigator, Allan Kaplan, Principle Investigator, Centre for Addiction and Mental Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 174/2010
Record Dates: First submitted 2017-04-24; First posted 2017-05-09 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Intervention Model Description: A pilot study to investigate the efficacy and safety of deep-rTMS delivered with the H-coil able to reach insula in subjects with long standing treatment resistant severe anorexia nervosa (TrAN)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Deep insula-coil rTMS (Experimental): Active treatment phase consists of deep rTMS (18 Hz, 2 sec on, 20 sec off, over approximately 30 min) 5 times per week, for 6 weeks, for a total of 30 sessions as a part of an active treatment phase.
  Maintaince treatment phase includes two sessions of rTMS (18 Hz, 2 sec on, 20 sec off, over approximately half an hour) weekly for the period of 6 weeks.
  Interventions: Device: Deep Insula-coil rTMS

INTERVENTIONS:
Device: Deep Insula-coil rTMS — Before administering TMS participants will undergo cue stimuli provocation, consisting of 32 professional color images of high calorie, sweet and savory food. This will follow with TMS. All subjects will receive prefrontal deep TMS (18 Hz, 2 sec on, 20 sec off, over approximately 30 min) 5 times per week, for 6 weeks, for a total of 30 sessions as a part of an active treatment phase. Maintenance treatment phase will include two sessions of rTMS (18 Hz, 2 sec on, 20 sec off, over approximately half an hour) weekly for the period of 6 weeks.
  Other Names: deep H-coil rTMS; deep insula rTMS

SUMMARY:
OBJECTIVE: Anorexia Nervosa (AN) is a complex disorder of unknown etiology that is characterized by disordered eating behaviors and specific psychopathology. In the course of anorexia around 50% will recover in the first 10 years, 25% will continue to experience symptoms but will be able to function, and 25% will go to develop chronic course, and by definition become severe treatment resistant(Tr). There is little if anything to offer to this population where the range of treatment options is limited to weight restoration interventions. Transcranial magnetic stimulation (rTMS) is a non-invasive intervention, which presents a particular interest in people with severe TrAN, specifically because of its ability to target deeper areas of the brain, such as insula, which has been argued to be a possible trait marker for AN. METHODS: This pilot study will test the efficacy and safety of deep-rTMS delivered with the H-coil in subjects with long standing treatment resistant severe anorexia nervosa (TrAN).

DETAILED DESCRIPTION:
Anorexia Nervosa (AN) is a complex disorder that is characterized by disordered eating behaviors and specific psychopathology. It is frequently unremitting, and is associated with significant morbidity and mortality. There are no effective evidenced based treatments for adult individuals who suffer from this disease, and innovative treatment strategies are constantly being sought. One potential novel treatment approach is brain stimulation, specifically repetitive transcranial magnetic stimulation (rTMS) which has been used to treat various neurobehavioural disorders, including anxiety and depression. There are a number of deep brain regions implicated in the etiology of AN, including the insula. The insula has been identified as an important region in AN pathophysiology. The insula has a role in gustatory modulation and feeding behavior, as well as the processing of interoceptive stimuli and self awareness. In a metanalysis of published fMRI studies in patients with anorexia nervosa, we found hyperactivity in the region of the insula. However activation of such deeper regions with TMS has to date been unachievable as TMS technology has not yet had the capacity to target such deep brain structures. The Brainsway H-coil reaches deep subcortical structures such as the insula.

This pilot study will investigate the efficacy and safety of the Brainsway H-coil deep brain rTMS in the treatment of patients with treatment resistant anorexia nervosa (TrAN). The general objective of this study is to investigate the neurological pathways implicated in AN using Hcoil deep rTMS. The specific goal is to test the safety and tolerability of repeated H-coil TMS as a potential treatment for TrAN. Also, if the safety and tolerability of deep H-coil rTMS stimulation is demonstrated in this study, this modality may be useful as a potential treatment strategy for individuals with AN. If both efficacy and safety are demonstrated, then a properly designed randomized controlled trial with deep H-coil rTMS compared to sham rTMS treatment will be implemented to investigate the possible therapeutic effects of H-Coil deep rTMS stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AN according to DSM-IV criteria: For DSM-IV, amenorrhea will not be strictly applied, as these subjects have been shown to be clinically indistinguishable from those with full criteria AN.
* Body Mass Index (BMI) > 14.0 kg/m2 and < 18.5 kg/m2
* Ages > 18 years, < 55 years
* Patient have had > 2 failed attempts at intensive nutritional rehabilitation, either in an inpatient or day hospital setting, and have been ill with AN for more than 5 years
* Medically stable
* Competent to provide Informed Consent
* Speak and understand English
* Safety Screening for rTMS (see exclusion criteria)

Exclusion Criteria:

* Any medical or psychiatric problem requiring urgent medical or psychiatric attention (e.g. acute suicidality),
* significant metabolic disturbance upon psychiatrist presentation (e.g., K+ < 2.5 mEq/L),
* patients with significant co-morbid illnesses that are not likely to benefit from proposed treatments or that need specialized treatments for non-eating disorder symptoms. (Note that once a participant is already in the study, participant may remain if medical problems develop but are corrected in a timely fashion. Please see criteria for study withdrawal for details)
* Pregnancy
* QTc > 480 msec at baseline or increase in QTc of > 35 msec since baseline ECG
* Significant systemic or metabolic illness; i.e.,diabetes mellitus( fasting blood sugar > 120 mg/dL or non-fasting > 140 md/dL) or hyperlipidemia ( cholesterol, triglycerides > 1.5 x upper limit of normal)
* Current diagnosis of substance abuse or dependence in past 6 months
* Diagnosis of schizophrenia, schizophreniform disorder, bipolar illness (type I)
* Significant neurological disorder, including past history of documented seizure, familial or personal history of epilepsy, ECT within past 3months prior to screening, history of rTMS in the past 3months
* Presence of any intracranial medical device, or any metal objects which may be present in the body
* Taking mood stabilizers or anticonvulsants. Subjects will be allowed in the study if they are taking a low stable dose of antidepressant or antipsychotic medication for a period of > 4 weeks at an unchanged dose.
* Participation in a psychotherapeutic intervention instituted within 3 months of the beginning of the trial. Subjects in psychotherapy at a stable frequency for at least the last 3 months prior to entering the study will be allowed to participate

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Seizures | bi-weekly through for 12 weeks
  absence of seizures as observed by clinical team and reported by participants

SECONDARY OUTCOMES:
Decrease in binge eating and purging in B/P group | b-weekly for 12 weeks
  as reported by participants
Increase in calorie intake | bi-weekly for 12 weeks
  as measured by self-report thorough the use of food journal
Decrease in depressive and anxiety | bi-weekly for 12 weeks
  as measured by HAMD, MADRS, BDI, and BDS
Decrease in AN-related obsessions and compulsions | bi-weekly for 12 weeks
  as measured by YBOCS-ED

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Blumberger, MD, FRCP(C), Study Chair — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No